CLINICAL TRIAL: NCT04171232
Title: Effect of Augmented Reality Intervention on the Range of Motion, Muscle Strength, Function of Upper Extremity and Balance in Children With Spastic Hemiplegic Cerebral Palsy: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zohra Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1402-ZIHS-013
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: Spastic; Hemiplegia; Cerebral palsy; Child; Upper Extremity; Range of Motion; Muscle Strength; Function; Balance; Augmented Reality; Intervention
MeSH Terms: conditions — Muscle Spasticity; Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Balance It (Group 1) (Active Comparator): Children with spastic hemiplegic cerebral palsy were assessed by Manual Muscle Testing (MMT) to determine the muscle power/strength, Goniometer to determine the Range of Motion (ROM), Disability of Arms, Shoulders, and Hand (DASH) questionnaire to assess the function of upper extremity, and Pediatric Balance Scale to determine the body balance and were assigned in the Balance It group. Each subject in first group would complete 8 weeks of augmented reality(AR) therapy sessions which would be aimed to improve the muscle power/strength, range of motion, balance and function. Each subject would be evaluated before their first AR therapy session (pre- interventionally) and after their last AR therapy session (post-interventionally) for changes in muscle power, ROM, upper extremity function and balance.
  Interventions: Other: Balance It
- Bubble Pop (Group 2) (Active Comparator): Children with hemiplegic cerebral palsy were assessed by Manual Muscle Testing (MMT) to determine the muscle power/strength, Goniometer to determine the Range of Motion (ROM), Disability of Arms, Shoulders, and Hand (DASH) questionnaire to assess the function of upper extremity, and Pediatric Balance Scale to determine the body balance and were assigned in the Bubble Pop group. Each subject in second group would complete 8 weeks of augmented reality(AR) therapy sessions which would be aimed to improve the muscle power/strength, range of motion, balance and function. . Each subject would be evaluated before their first AR therapy session (pre- interventionally) and after their last AR therapy session (post-interventionally) for changes in muscle power, ROM, upper extremity function and balance.
  Interventions: Other: Bubble Pop
- Scoop'd (Group 3) (Active Comparator): Children with hemiplegic cerebral palsy were assessed by Manual Muscle Testing (MMT) to determine the muscle power/strength, Goniometer to determine the Range of Motion (ROM), Disability of Arms, Shoulders, and Hand (DASH) questionnaire to assess the function of upper extremity, and Pediatric Balance Scale to determine the body balance and were assigned in the Scoop'd group. Each subject in third group would complete 8 weeks of augmented reality(AR) therapy sessions which would be aimed to improve the muscle power/strength, range of motion, balance and function. . Each subject would be evaluated before their first AR therapy session (pre- interventionally) and after their last AR therapy session (post-interventionally) for changes in muscle power, ROM, upper extremity function and balance
  Interventions: Other: Scoop'd

INTERVENTIONS:
Other: Balance It — Each patient in group 1 i.e. Balance It group would be given a 15 minutes long session. Each session would start in standing position and the patient would play the game while they would be instructed to balance the objects falling from above on the imaginary bar (and an actual bar at later stages) held with their both hands, and not let those objects fall by opening their arms wide open and by staying or moving according to the target spot for the set time. This session would be repeated three times a week for two months (total 12 sessions/month).
  Arms: Balance It (Group 1)
Other: Bubble Pop — Each patient in group II i.e. Bubble Pop group would be given a 15 minutes long session. Each session would start in standing position and the patient would play the game while they would be instructed to reach for the balloons coming from random directions and pop them by moving their upper limbs and even their whole body if required. They would also be instructed to avoid a specific object that would result in deduction of their overall game score. This session would be repeated three times a week for two months (total 12 sessions/month).
  Arms: Bubble Pop (Group 2)
Other: Scoop'd — Each patient in group III i.e. Scoop'd group would be given a 15 minutes long session. Each session would start in standing position and the patient would play the game while they would be instructed to hold an imaginary ice cream cone (and an actual basket designed similar to an ice cream cone in later stages) with their both hands and move to catch the ice cream scoops falling at random spots from above, one spot at a time. They would also be instructed to avoid a specific object that would result in deduction of their overall game score. This session would be repeated three times a week for two months (total 12 sessions/month).
  Arms: Scoop'd (Group 3)

SUMMARY:
Cerebral Palsy (CP) is a disorder of the development of movement and posture, causing activity limitations attributed to nonprogressive disturbances of the fetal or infant brain that may also affect sensation, perception, cognition, communication, and behavior. Motor control during reaching, grasping, and walking are disturbed by spasticity, dyskinesia, hyperreflexia, excessive coactivation of antagonist muscles, retained developmental reactions, and secondary musculoskeletal malformations, together with paresis and defective programing. Weakness and hypoextensibility of the muscles are due not only to inadequate recruitment of motor units, but also to changes in mechanical stresses and hormonal factors. As it affects the children, therefore it should be emphasized. Effect of Augmented Reality (AR) based therapeutic games on the range of motion, muscle strength,function of upper limb and balance of spastic hemiplegic cerebral palsy children would be assessed through goniometer, manual muscle testing (MMT), disability of Arms, Shoulders, and Hand (DASH) questionnaire, and Pediatric Berg Balance Scale, respectively.

DETAILED DESCRIPTION:
A total of 30 children with spastic hemiplegic cerebral palsy would be recruited and randomly divided into three groups, 10 in each group. The demo-graphical data would be collected through a general demographic questionnaire. Outcome measures would include Goniometer to determine the Range of Motion (ROM), Manual Muscle Testing (MMT) to determine the upper limb muscle power/strength, disability of Arms, Shoulders, and Hand (DASH) questionnaire to assess the function of upper extremity, and Pediatric Balance Scale to determine the body balance.

ELIGIBILITY:
Inclusion Criteria:

Children with diagnosed spastic hemiplegic cerebral palsy, aged between 6 to 12 years, having sufficient cognitive capacity to understand the basic instructions and to cooperate with the instructor during the assessment and intervention, ambulant- classified as level 1 or 2 on Gross Motor Functional Classification System, able to move the affected body parts easily, and sufficient for functional activity- score of 1 or 2 on Modified Ashworth Scale, good general health, without any other known neurological or orthopedic diagnoses, as confirmed by health professionals and their parents.

Exclusion criteria:

Children who have received motor therapy treatment (e.g. Botulinum Toxin/Constraint-Induced Movement Therapy) in the past six months or plan to receive such treatment during the study,those with severe attention deficits, or those who have a history of seizures which can be triggered by television light (confirmed by the child's therapist or pediatric neurologist), or those children who have visual and/or hearing impairments, or children with musculoskeletal contractures or deformities will be excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Testing | Upto 8 weeks
  Muscle power would be measured through Manual Muscle Testing with categories as:
  Grade 0= No evidence of contractility (complete paralysis) Grade 1= Slight contractility without any movement Grade 2= The patient completes full or partial range of motion with gravity eliminated Grade 3= Completes the available test range of motion against gravity, but tolerates no resistance Grade 4= Movement against gravity plus some resistance Grade 5= Movement against gravity plus full resistance
Goniometer | Upto 8 weeks
  Range of motion would be measured through Goniometer
Pediatric Balance Scale | Upto 8 weeks
  Body balance would be assessed through Pediatric Balance Scale
Disability of Arms, Shoulders and Hand Questionnaire (DASH) | Upto 8 weeks
  Disability of Arms, Shoulders and Hand Questionnaire (DASH) would be used to assess the upper limbs' function

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Rehabilitation Medicine, Islamabad, Punjab, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- [Derived] Malick WH, Butt R, Awan WA, Ashfaq M, Mahmood Q. Effects of Augmented Reality Intervention on the Range of Motion and Muscle Strength of Upper Extremity in Children with Spastic Hemiplegic Cerebral Palsy: A Randomized Clinical Trial. Games Health J. 2022 Jun;11(3):168-176. doi: 10.1089/g4h.2021.0128. Epub 2022 Mar 14. PMID 35285674